CLINICAL TRIAL: NCT01110070
Title: Pivotal Study in Europe for CE Mark
Brief Title: ChonDux for Filling Full Thickness Cartilage Defects in the Femoral Condyle of the Knee
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment suspended; follow up continue
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCS-08
Record Dates: First submitted 2010-04-22; First posted 2010-04-26 (Estimated); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Cartilage Defect
Keywords: articular; cartilage; microfracture; knee pain; cartilage repair; Subjects with an articular cartilage defect in the knee.
MeSH Terms: conditions — Fractures, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ChonDux plus microfracture (Experimental)
  Interventions: Device: ChonDux
- Microfracture (Active Comparator)
  Interventions: Device: ChonDux

INTERVENTIONS:
Device: ChonDux — Comparison of ChonDux plus microfracture to microfracture only
Device: ChonDux — single use device
  Arms: Microfracture

SUMMARY:
The use of ChonDux Cartilage Repair system for the treatment of single cartilage lesions in the femoral condyle of the knee. The primary outcome measure is degree of lesion fill at 6 months. Filling of the femoral chondral defect of the knee using ChonDux™ Cartilage System may give symptomatic relief of pain and help to restore knee function. Included in this study is pain relief using Visual Analog Scale (VAS), knee function using the International Knee Documentation Committee (IKDC) questionnaire and quality of life using the Short Form-36 (SF-36) survey.

DETAILED DESCRIPTION:
Current treatment approaches for articular cartilage defects have been disappointing and clinical results have been variable. However, when using crosslinked hydrogel technologies, in vitro findings have shown chondrocyte growth and extra-cellular matrix (ECM) production supportive of cartilage production.

ELIGIBILITY:
Inclusion Criteria:

* A standing radiograph of the knee showing a Kellgren score of 0-2
* Body mass index ≤33
* An Outerbridge score of III or IV without need for bone graft
* A meniscus with no more than partial resection in the affected knee

Exclusion Criteria:

* Passive motion deficit of the knee (>5º of extension, >15º of flexion)
* Moderate or severe osteoarthritis
* Diabetes mellitus (IDDM Type 1)
* Patellofemoral instability
* Malalignment with > 5° valgus or varus compared to contralateral knee
* Active osteomyelitis

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2010-07; Primary Completion 2010-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Defect fill at 6 months determined by magnetic resonance imaging (MRI) | 6 months

SECONDARY OUTCOMES:
Pain score (VAS) | 6 months
Knee function as assessed by the IKDC questionnaire | 6 months
SF-36 Health Survey | 6 months

CONTACTS AND LOCATIONS:
Locations (7):
- Austria (2):
  - Medalp, Imst
  - Ortho.Abteilung, AKH Linz, Linz
- Germany (3):
  - Krakenhaus Altentreptow, Altentreptow
  - Orthopedic and Pain Center Freiberg, Freiberg
  - University Mannheim, Mannheim
- Netherlands (2):
  - Meander Medical Center, Baarn
  - Tergooiziekenhuizen, Hilversum

REFERENCES:
- [Derived] Wolf MT, Zhang H, Sharma B, Marcus NA, Pietzner U, Fickert S, Lueth A, Albers GHR, Elisseeff JH. Two-Year Follow-Up and Remodeling Kinetics of ChonDux Hydrogel for Full-Thickness Cartilage Defect Repair in the Knee. Cartilage. 2020 Oct;11(4):447-457. doi: 10.1177/1947603518800547. Epub 2018 Oct 3. PMID 30280586